CLINICAL TRIAL: NCT00348101
Title: The Influence of Continuous Perioperative Beta-Blocker Therapy in Combination With Phosphodiesterase Inhibition on Cardiac Neurohormonal Activation and Myocardial Ischaemia in High-Risk Vascular Surgery Patients
Brief Title: Effects of Beta-Blocker Therapy and Phosphodiesterase Inhibition on Cardiac Neurohormonal Activation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Klinikum Ludwigshafen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESPEKLILU05
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-04

CONDITIONS: Coronary Artery Disease
Keywords: Patients undergoing major vascular surgery having documented CAD or risk factors for CAD
MeSH Terms: conditions — Coronary Artery Disease | interventions — Psychotherapy, Multiple; Enoximone; esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Combined therapy with enoximone and esmolol

SUMMARY:
Previous clinical investigations have demonstrated the utility of β-adrenergic blockade in reducing perioperative ischaemic events, ultimately translating into a decrease in cardiac morbidity and mortality. However, β-blocker therapy remains underutilized in clinical practice because of concerns of potential adverse effects such as a reduced inotropic state, which might result in acute congestive heart failure or hypotension. Therefore, additional treatment with a positive inotropic agent might be needed. Phosphodiesterase inhibitors (PDEIs) offer a favourable pharmacological profile in this setting and stimulate cardiac function in the absence of the β-adrenergic receptor.

We hypothesize that the combination of PDEI and β-blocker therapy would decrease perioperative plasma concentrations of brain natriuretic peptide (BNP) in patients requiring major vascular surgery. BNP is chosen as our primary outcome variable because of its importance as a sensitive correlate of myocardial dysfunction and its prognostic value for predicting the risk of cardiac death across the entire spectrum of acute coronary syndromes.

DETAILED DESCRIPTION:
Cardiac complications, such as, myocardial infarction, heart failure, and life-threatening dysrhythmias, are the leading cause of perioperative death among patients undergoing major vascular surgery.

The pathogenesis of perioperative ischaemic events is most certainly multifactorial and includes persistent activation of several neurohormonal pathways, such as the natriuretic peptide system.

Previous clinical investigations have demonstrated the utility of β-adrenergic blockade in reducing perioperative ischaemic events, ultimately translating into a decrease in cardiac morbidity and mortality especially in patients who had or were at high risk for coronary artery disease. Therefore, the administration of β-blockers to all patients at high risk for coronary events who are scheduled to undergo major noncardiac surgery is strongly supported by consensus recommendations and clinical guidelines. Despite the evidence of benefit, β-blockers remain underutilized in clinical practice because of concerns of potential adverse effects such as a reduced inotropic state, which might result in myocardial depression, acute congestive heart failure, and hypotension [13]. Therefore, additional treatment with a positive inotropic agent might be needed.

Phosphodiesterase inhibitors (PDEIs) offer a favourable pharmacological profile in this setting and retain their haemodynamic effects in the face of full β-blockade. Preliminary data suggest that the combination of PDEI and β-blocker therapy may be better tolerated and allows for expression of the known effects of β-blocker therapy and improved myocardial functioning without the adverse effects of either therapy alone.

We therefore hypothesize that the combination of PDEI and β-blocker therapy would decrease perioperative plasma concentrations of brain natriuretic peptide (BNP) in patients requiring major vascular surgery documented to have a high prevalence of coronary artery disease and limited coronary reserve. BNP is chosen because of its pivotal role as a sensitive correlate of myocardial dysfunction and its prognostic value for predicting the short- and long-term risk of cardiac death across the entire spectrum of acute coronary syndromes.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for major vascular surgery
* can sign informed consent before surgery
* documented CAD or risk factors for CAD

Exclusion Criteria:

* Preoperative treatment with beta-adrenergic agonists or glucocorticoids,
* electrocardiographic (ECG) abnormalities like nonsinus rhythm, second- or third degree heart block, or left bundle branch block,
* cardiac pacemaker dependency,
* symptomatic mitral or aortic valvular disease,
* a history of asthma, bronchospasm, or severe chronic obstructive pulmonary disease necessitating bronchodilator therapy,
* severe liver dysfunction
* known allergies against the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-06; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
We hypothesize that the combination of PDEI and β-blocker therapy
would decrease perioperative plasma concentrations of brain natriuretic peptide
BNP) in patients requiring major vascular surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Suttner, M.D., Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine Klinikum Ludwigshafen, Ludwigshafen, Germany

REFERENCES:
- [Derived] Suttner S, Boldt J, Mengistu A, Lang K, Mayer J. Influence of continuous perioperative beta-blockade in combination with phosphodiesterase inhibition on haemodynamics and myocardial ischaemia in high-risk vascular surgery patients. Br J Anaesth. 2009 May;102(5):597-607. doi: 10.1093/bja/aep062. Epub 2009 Mar 31. PMID 19336536 (Retraction: PMID 21685126 Reilly C. Br J Anaesth. 2011 Jul;107(1):116-7)